CLINICAL TRIAL: NCT05030415
Title: A Proof of Concept, Non-randomized, One Center Study to Explore the Safety and Efficacy of 16 Weeks of Treatment With Ixekizumab in Adult Patients With Lichen Planus and Lichen Planopilaris
Brief Title: Ixekizumab in Adult Patients With Lichen Planus and Lichen Planopilaris
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, John R. Durkin, Assistnat Professor of Dermatology, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-087
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Lichen Planus Scalp; Lichen Planus; Lichen Planopilaris
Keywords: IL17 lichen planus
MeSH Terms: conditions — Lichen Planus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ixekizumab (Experimental): ixekizumab 80 mg injection, 160 mgs injected subcutaneously on week 0, 80 mgs injected subcutaneously every two weeks
  Interventions: Drug: Ixekizumab Auto-Injector

INTERVENTIONS:
Drug: Ixekizumab Auto-Injector — 160 mg week 0 followed by 80 mg every two weeks

SUMMARY:
To evaluate the safety and efficacy of ixekizumab in lichen planus and lichen planopilaris clinical response by Total Body Surface (TBS) determination, Investigator Global Assessment (IGA) Score, Lichen Planopilaris Activity Index (LPPAI), and Frontal Fibrosing Alopecia Severity Score (FFASS).

DETAILED DESCRIPTION:
A proof of concept, non-randomized, one center study to explore the safety and efficacy of 16 weeks of treatment with ixekizumab in adult patients with lichen planus. The total study period will consist of 24 weeks including a 2 week screening/washout, 16 weeks of active therapy and 8 weeks of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for study participation must be obtained before any study assessment is performed
* Male and female patients 18 years or older at the time of screening
* Patients who are willing and capable of cooperating to the extent and degree required by the protocol
* Patients who read and sign an approved informed consent for this study
* Clinical diagnosis of cutaneous lichen planus, lichen planopilaris, frontal fibrosing alopecia at least 6 months prior to enrollment as determined by patient interview of his/her medical history, biopsy proven lichen planus and by confirmation of diagnosis through physical examination by the investigator
* Failure to at least one topical treatment (including but not exclusively topical corticosteroids, topical calcineurin inhibitors, topical vitamin D analogues) and/or systemic treatments (including but not exclusively systemic retinoids, griseofulvin, sulfasalazine, hydroxychloroquine, light therapy, methotrexate, etc.) for 4 weeks

Exclusion Criteria:

* Forms of diagnosed lichen planus other than cutaneous or lichen planopilaris
* Previous exposure to ixekizumab or any other biologic drug directly targeting IL-17A or IL-17RA receptors (e.g., secukinumab, brodalumab, etc)
* Presence of skin comorbidities that may interfere with study assessments
* Plans for administration of live vaccines during the study period or within 6 weeks before randomization
* Use of any investigational treatment within 4 weeks prior to Randomization, or within a period of 5 half-lives of the investigational treatment prior to Randomization, whichever is longer
* Currently enrolled in any other clinical trial involving any investigational agent or device
* Known history of positive hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody. If a patient has a documented negative result for any of these tests within 1 year of baseline, that particular test is not required at screening. Patients with isolated positive HBcAb or with positive hepatitis C antibody may undergo additional tests and consultations, and may enter the study only if active hepatitis B infection or carrier status has been definitively ruled out
* Known history of human immunodeficiency virus (HIV) infection or HIV seropositivity (HIV testing is not required at screening for patients with a negative HIV result within the past 1 year prior to baseline)
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for skin Bowen's disease, non-invasive squamous cell carcinoma, basal cell carcinoma, actinic keratosis that have been treated, carcinoma in situ of the cervix, or non-invasive malignant colon polyps that have been removed)
* History or evidence of ongoing alcohol or drug abuse, within the last 6 months prior to randomization
* History of elevated liver functioning tests 2-3 times of its normal
* Current requirement for systemic immunosuppressive/ immunomodulatory agent (including but not exclusively metronidazole) other than study Ixekizumab; if currently on immunosuppressive/ immunomodulatory therapy, excluded if not possible to have washout period of 2 weeks for topicals and 4 weeks for systemic required
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study. Examples include, but are not limited to patients with short life expectancy, patients with uncontrolled diabetes (HbA1c ≥9%), patients with cardiovascular conditions (eg, stage III or IV cardiac failure according to the New York Heart Association classification), severe renal conditions (eg, patients on dialysis), neurological conditions (eg, demyelinating diseases), active major autoimmune diseases (eg, lupus, inflammatory bowel disease, rheumatoid arthritis, etc.), other severe endocrinological, gastrointestinal, hepato-biliary, metabolic, pulmonary or lymphatic diseases. The specific justification for patients excluded under this criterion will be noted in study documents
* Any other medical or psychological condition (including relevant laboratory abnormalities at screening) that, in the opinion of the investigator, may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study patient as a result of his/her participation in this clinical trial, may make patient's participation unreliable, or may interfere with study assessments. The specific justification for patients excluded under this criterion will be noted in study documents
* Active systemic infections during 2 weeks prior to randomization (exception: the common cold) or any infection that reoccurs on a regular basis
* History of an ongoing, chronic or recurrent infectious disease, or positive or indeterminate QuantiFERON TB-Gold test at screening
* Planned major surgical procedure during the patient's participation in this study
* Patient is a member of the investigational team or his/her immediate family
* Pregnant or nursing women; women planning a pregnancy within the study period
* Women unwilling to use adequate birth control, if of reproductive potential* and sexually active. Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception whenever engaging in heterosexual intercourse throughout the duration of the study and for 16 weeks after last dose of study drug. These include: hormonal contraceptives, intrauterine device (IUD), a double barrier method (eg, condom + diaphragm), or male partner with documented vasectomy.

  * For females, menopause is defined as at least 12 consecutive months without menses; if in question, a follicle stimulating hormone (FSH) of ≥25 mU/mL must be documented. Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable; if documented, women with these conditions are not required to use additional contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment (IGA) | 16 weeks
  Change in IGA

SECONDARY OUTCOMES:
Lichen Planopilaris Activity Index (LPPAI) | 16 weeks
  Change in LPPAI
Frontal Fibrosing Alopecia Severity Score (FFASS) | 16 weeks
  Change in FFASS

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monteiro BV, Pereira Jdos S, Nonaka CF, Godoy GP, da Silveira EJ, Miguel MC. Immunoexpression of Th17-related cytokines in oral lichen planus. Appl Immunohistochem Mol Morphol. 2015 Jul;23(6):409-15. doi: 10.1097/PAI.0000000000000096. PMID 25356945